CLINICAL TRIAL: NCT03764839
Title: "My Surgical Success": A Randomized Controlled Trial of a Perioperative Digital Behavioral Pain Medicine Treatment Tested in Orthopedic Trauma Patients
Brief Title: Digital Behavioral Pain Medicine for Orthopedic Trauma Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Beth Darnall, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42569
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Orthopedic Trauma Surgery Patients
Keywords: pain; treatment; opioid cessation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control Group (Digital Health Education) (No Intervention): * Demographics survey
  * Baseline surveys
  * Participants receive a digital information sheet on nutrition and exercise that are relevant for people recovering from surgery. Participants are encouraged to incorporate healthy lifestyle choices into their daily routines as they recover from surgery
  Post-surgery:
  * Pain check-ins (2 times per week) (detailed above)
  * Patients receive 30 second booster videos at 7, 14, and 21 days after surgery
  * Follow-up surveys (4, 8, and 12 weeks after surgery)
- "My Surgical Success" Treatment Group (Experimental): * Demographics survey
  * Baseline surveys
  * Intervention:
    * 45-minute digital behavioral pain medicine intervention "My Surgical Success" that emphasized cognitive and emotional regulation of pain and downregulation of physiologic arousal.
    * downloadable app with an audio file
    * personalized plan that allows learners to incorporate the treatment information
  * Post-video survey (detailed above)
  Post-surgery:
  * Pain check-ins (2 times per week) (detailed above)
  * Follow-up surveys (4, 8, and 12 weeks after surgery) Intervention: Behavioral: Perioperative Digital Behavioral Pain Medicine "My Surgical Success"
  Interventions: Behavioral: Perioperative Digital Behavioral Pian Medicine "My Surgical Success"

INTERVENTIONS:
Behavioral: Perioperative Digital Behavioral Pian Medicine "My Surgical Success" — The "My Surgical Success" website include 45 minutes of psychoeducation material developed and delivered by Beth Darnall, PhD. Viewers learn basic skills to improve regulation of pain-related distress. Treatment includes an app and a personalized plan for surgical success.
  Arms: "My Surgical Success" Treatment Group

SUMMARY:
The primary purpose of this study is to determine the feasibility and preliminary efficacy of a perioperative digital behavioral pain medicine intervention delivered to orthopedic trauma surgery patients (compared to an active control group that receives digital health education).

Aim 1: Determine feasibility of and satisfaction, and perceived utility of "My Surgical Success"

Hypothesis 1: For My Surgical Success, the investigators anticipate 50% engagement in the study (feasibility). Of those who complete My Surgical Success, the investigators expect 80% satisfaction ratings, and 80% perceived utility of the information learned.

Aim 2: Determine group differences in time to post-surgical pain and opioid cessation.

Hypothesis 2: "My Surgical Success" participants will evidence quicker time to post-surgical pain and opioid cessation compared to the HE Control Group.

Aim 3: Determine group differences in within-subject pain catastrophizing scores (baseline to post-surgery).

Hypothesis 3: "My Surgical Success" participants evidence greater reduction in pain catastrophizing (measured with the Pain Catastrophizing Scale; PCS) compared to the HE Control group.

Aim 4: Determine group differences in post-surgical psychological correlates (PROMIS Depression, Anxiety, Function, Pain Interference, Sleep Disturbance, Social Isolation, Fatigue, and Pain Intensity).

Hypothesis 4: "My Surgical Success" participants will evidence greater post-surgical function and lower pain related interference compared to the HE Control Group.

The goal of this research is to advance our understanding regarding the feasibility and effectiveness of "My Surgical Success" (a digital, perioperative behavioral pain medicine treatment) and its impact on post-surgical outcomes.

DETAILED DESCRIPTION:
Patients are identified by their orthopedic surgeon or study personnel immediately prior to surgery or during their stay on the inpatient post-surgical recovery unit. Beyond recruitment, the entire study is conducted remotely with no in-person contact with study staff. After enrollment, study staff follow-up with patients by phone, text or email (depending on patient preference); informed consent is obtained online.

All participants are asked to provide baseline demographic information, as well as self-reported measures assessing mood, pain, cognitive and emotional responses to pain, catastrophizing, and medications. All measures are administered via a secure, HIPAA compliant, online system (REDCap).

Participants are then randomized to receive one of two digital treatments: a behavioral pain medicine intervention ("My Surgical Success") or to a health education (HE Control). Participants who have been randomized to the HE control group receive online text information about health and nutrition, and are oriented that the information is relevant for improving recovery from surgery. The digital behavioral pain medicine intervention emphasizes treatment content that targets cognitive and emotional regulation in the context of pain. "My Surgical Success" includes three brief psychoeducational video learning modules, a downloadable app with an audio file, and a downloadable PDF Personalized Plan for Success. After participants in the "My Surgical Success" group view the online treatment videos, they complete questions regarding their satisfaction with the video content, perceived usefulness of information, and likelihood to use the skills learned. All participants are tracked twice per week post-surgically to assess pain and opioid use. Data are captured for the duration of the study (12 weeks) or until patients reach opioid cessation (four consecutive surveys indicating zero opioid use). Psychosocial data are collected post-surgically at weeks 4, 8, and 12.

Post-treatment questions:

Participants in the "My Surgical Success" group are asked to rate questions about the about the video content in regards to its understandability, relevance, usefulness, their overall satisfaction, how likely they are to use the information learned.

Following surgery, all participants fill out online brief pain check-ins (2 times per week) to assess pain and medication use. Daily measures continue until the participant reports 4 consecutive reports of zero opiate use. Until reaching this endpoint, pain check-ins are collected for 12 weeks (the duration of the study).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Undergoing a scheduled surgery for orthopedic trauma
* Post-surgery up to 7 days
* English fluency
* Ability and willingness to complete electronic study procedures including questionnaires, assessments, and receipt of treatment.

Exclusion Criteria:

* Any conditions causing inability to complete study procedures (e.g. cognitive ability, mental status, medical status) or lack of access to internet and phone that would prevent participation in study procedures - at the discretion of the staff member.
* long-term opioid use prior to surgery
* Known pregnancy
* Ongoing legal action related to pain or disability claim
* Multiple surgeries and/or infections
* Injury is not fracture related or non-trauma surgery
* Documented history of alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
Participant ratings (0-6) for acceptability, satisfaction, usefulness of the information presented, ease of understanding, and likelihood to use skills learning (for the My Surgical Success group only) | Immediately post-treatment
  Participants complete a single time point rating for 5 items listed above. Ratings occur on a 0-6 point scale (e.g., 0=completely useless and 6=Very useful). Percentages will be reported for each item. A higher score indicates better acceptability, satisfaction, usefulness of the information.
Group difference in time to pain and opioid cessation | This is a survival curve with time being a variable of interest. The examination will occur within the 3-month window after surgery.
  This will be measured in days until patients achieve opioid cessation. Fewer days indicate better treatment effects

SECONDARY OUTCOMES:
Group difference in within-subject Pain Catastrophizing Scale (PCS) | Baseline to 1 month
  PCS measures pain catastrophizing

OTHER OUTCOMES:
Group differences in post-surgical Patient Reported Outcomes Measurement Information System (PROMIS) function and PROMIS average pain intensity | Post-surgical month 1
  PROMIS function measures patients' level of physical functioning, and PROMIS pain intensity measures patients' average level of pain intensity. PROMIS scores for function and pain interference will be reported at month 1. The investigators will conduct within subject analyses and will report pre-post treatment changes. Also, the investigators will aggregate scores by group and conduct between group analyses to report differences between group means and SD. Higher value on PROMIS function indicates better levels of physical functioning and higher levels of PROMIS pain intensity indicate worse pain levels.
Characterize responders to "My Surgical Success" (demographics and psychological correlates) | Baseline
  The investigators with report the baseline demographic and psychosocial scores for patients who report high satisfaction with the "My Surgical Success" treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ziadni MS, You DS, Keane R, Salazar B, Jaros S, Ram J, Roy A, Tanner N, Salmasi V, Gardner M, Darnall BD. "My Surgical Success": Feasibility and Impact of a Single-Session Digital Behavioral Pain Medicine Intervention on Pain Intensity, Pain Catastrophizing, and Time to Opioid Cessation After Orthopedic Trauma Surgery-A Randomized Trial. Anesth Analg. 2022 Aug 1;135(2):394-405. doi: 10.1213/ANE.0000000000006088. Epub 2022 Jul 5. PMID 35696706